CLINICAL TRIAL: NCT06624098
Title: Early Transjugular Intrahepatic Portosystemic Shunt for Advanced Hepatocellular Carcinoma With Main Trunk Portal Vein Tumor Thrombus Induced Gastrointestinal Bleeding: a Multicenter Phase II Study
Brief Title: Early Transjugular Intrahepatic Portosystemic Shunt for Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Zhou Qunfang, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Liver Projiect 12
Record Dates: First submitted 2024-10-01; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Advanced Hepatocellular Carcinoma; Variceal Bleeding
Keywords: Advanced hepatocellular carcinoma; Variceal bleeding; Therapeutic endoscopy; Transjugular intrahepatic portosystemic shunt

STUDY DESIGN:
Intervention Model Description: Early transjugular intrahepatic portosystemic shunt (TIPS) within 72 hours after acute variceal bleeding.
Masking Description: TIPS was performed within 72 hours after variceal bleeding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early transjugular intrahepatic portosystemic shunt (TIPS) (Experimental): TIPS was performed within 72 hours after the endoscopic hemostasis.
  Interventions: Procedure: Early TIPS

INTERVENTIONS:
Procedure: Early TIPS — TIPS was performed within 72 hours after the endoscopic hemostasis.

SUMMARY:
Hepatocellular carcinoma (HCC) with main trunk portal vein tumor thrombus (PVTT) has poor prognosis. The main lethiferous factor is the upper gastrointestinal hemorrhage by PVTT-related portal hypertension. Studies have proven that early transjugular intrahepatic portosystemic shunt (TIPS) with 72 hours after acute variceal bleeding is effective.

DETAILED DESCRIPTION:
Portal hypertension by main trunk portal vein tumor thrombus (PVTT) is a severe disease. Patients usually die of gastrointestinal hemorrhage rather than tumor progression. It is vital to prevent the portal hypertension. Transjugular intrahepatic portosystemic shunt (TIPS) is an effective method to alleviate the portal pressure. Then the risk of gastrointestinal hemorrhage is decreased which provides an opportunity for system therapy. Studies have proven that early transjugular intrahepatic portosystemic shunt (TIPS) with 72 hours after acute variceal bleeding is effective for cirrhosis induced portal hypertension. However, the PVTT induced portal hypertension still needs clinical evidence. In this study, the investigators explore the early TIPS for advanced hepatocellular carcinoma with main trunk portal vein tumor thrombus induced acute variceal bleeding. The investigators aim to added clinical evidence for this subtype of advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of primary HCC, confirmed histologically or clinically according to the criteria of the American Association for the Study of Liver Diseases;
2. presence of PVTT with III-IV grade by Cheng's criteria;
3. having PVTT induced portal hypertension;
4. TIPS was performed within 72 hours after the endoscopic hemostasis;
5. metastases with limited five sites and no more two organs involved;
6. number of Intrahepatic tumors were no more than five;
7. receipt of Lenvatinib and PD-1 inhibitor as the first-line systemic therapy;
8. classified as Child-Pugh class A or B and having an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 2;
9. no history of other malignancies;
10. agreed to participated in this clinical trial;
11. Hemameba ≥3.0 x109/L, neutrophil ≥1.5x109/L, hemoglobin≥10.0 g/L, platelet≥100x 109/L, ALT; AST; bilirubin ≤1.5-fold normal, GFR≥60ml/min.

Exclusion Criteria:

1. recurrent HCC;
2. PVTT at I-II grade by Cheng's criteria;
3. age < 18 years or > 75 years;
4. advanced HCC with more than five metastases;
5. Number of Intrahepatic tumors were more than five;
6. no response to Lenvatinib;
7. life expectancy less than 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Rates of technical success | 3 months
  Patients did not occur gastrointestinal hemorrhage and the stent unobstructed 3 months after TIPS.

SECONDARY OUTCOMES:
Rates of gastrointestinal hemorrhage | 6 months
  Patients occur gastrointestinal hemorrhage within 6 months after TIPS.
Progression-Free-Survival (PFS) | 12 months
  Progression was defined as progressive disease by independent radiologic review.
Overall survival (OS) | 12 months
  OS is the length of time from the date of inclusion until death from any cause.
Objective response rate (ORR) | 12 months
  ORR, as determined based on tumor response according to RECIST 1.1, is defined as the proportion of all included patients whose best overall response (BOR) is either a complete response or partial response.
Adverse events | 12 months
  Safety will be evaluated according to the NCI CTCAE Version 4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Duan, MD, Study Director — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General hospital, Beijing, Beijing Municipality, China